CLINICAL TRIAL: NCT03611010
Title: Phase II, Dose-ranging Study to Evaluate the Efficacy Dose Response and Pharmacokinetics of Intravenous Atorvastatin in Hypercholesterolemic Patients Previously Controlled With Oral Atorvastatin
Brief Title: Dose-ranging Efficacy and Pharmacokinetics Study of Intravenous Atorvastatin in Hypercholesterolemic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CPI-1103-002
Record Dates: First submitted 2018-07-19; First posted 2018-08-02 (Actual); Results first posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-05

CONDITIONS: Hypercholesterolemia; Dyslipidemias
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias | interventions — Atorvastatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Cohort 1 = Baseline daily dose of 10 mg oral atorvastatin during lead-in, then IV study drug for up to 15 days
  Interventions: Drug: Atorvastatin injection
- Cohort 2 (Experimental): Cohort 2 = Baseline daily dose of 20 mg oral atorvastatin during lead-in, then IV study drug for up to 15 days
  Interventions: Drug: Atorvastatin injection
- Cohort 3 (Experimental): Cohort 3 = Baseline daily dose of 40 mg oral atorvastatin during lead-in, then IV study drug for up to 15 days
  Interventions: Drug: Atorvastatin injection
- Cohort 4 (Experimental): Cohort 4 = Baseline daily dose of 20 mg oral atorvastatin during lead-in, then SC study drug for up to 15 days
  Interventions: Drug: Atorvastatin injection

INTERVENTIONS:
Drug: Atorvastatin injection — statin (i.e., 3-hydroxy-3-methylglutaryl-coenzyme A (HMG-CoA) reductase inhibitor) for injection

SUMMARY:
Open-label study will titrate doses of intravenous atorvastatin and monitor respective LDL-C levels in hypercholesterolemic patients previously controlled on oral atorvastatin.

ELIGIBILITY:
Inclusion Criteria:

* On stable dose of daily oral atorvastatin for >= 5 weeks (oral atorvastatin may be provided during a lead-in period for subjects not previously taking atorvastatin)
* Stable LDL-C confirmed in the previous 7 to 10 days prior to enrollment into the treatment phase.

Exclusion Criteria:

* History of myopathy or rhabdomyolysis
* Liver disease including current biliary disorders
* Positive for HIV, Hepatitis B or Hepatitis C Virus
* Abuse of alcohol or non-prescribed drugs
* Unstable angina or arrhythmias or a cardiac event in the previous three months
* hypothyroidism, diabetes, or hypertension that is not under control
* pregnant or plans to be pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Tracey, MD, Principal Investigator — Frontage Lab
Locations (1):
- Frontage Clinical Services, Secaucus, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred between 07Aug2018 and 24Feb2020. Three types of patients, categorized by statin use prior to study participation were eligible: patients taking oral atorvastatin, patients taking statins other than atorvastatin, patient not taking any statins prior to study.
  In Amendment 03. the fourth 80mg dose was eliminated and the 15 days IV route administration was changed to subcutaneous administration.
Period: Period 1: Lead-In
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 14 | 14 | 2 | 10
Completed | 14 | 14 | 2 | 10
Not Completed | 0 | 0 | 0 | 0
Period: Period 2: 15 Day Treatment
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 14 | 14 | 2 | 10
Completed | 13 | 14 | 2 | 10
Not Completed | 1 | 0 | 0 | 0
Not completed — Inaccessible veins | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: All subjects who received at least a partial dose of investigational medicinal product. No treated subjects were excluded from the safety population.
Groups:
- Cohort 1: Cohort 1 = Baseline daily dose of 10 mg oral atorvastatin receiving either IV or SC study drug
- Cohort 2: Cohort 2 = Baseline daily dose of 20 mg oral atorvastatin receiving either IV or SC study drug
- Cohort 3: Cohort 3 = Baseline daily dose of 40 mg oral atorvastatin receiving either IV or SC study drug
- Cohort 4: Cohort 4 = Baseline daily dose of 20 mg oral atorvastatin receiving either SC study drug
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total
Number analyzed (Participants) | 14 | 14 | 2 | 10 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (9.74) | 51.4 (8.21) | 46.0 (18.38) | 50.4 (10.47) | 48.6 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 1 | 5 | 17
  Male | 8 | 9 | 1 | 5 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 1 | 4 | 17
  Not Hispanic or Latino | 7 | 9 | 1 | 6 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 6 | 0 | 4 | 15
  White | 9 | 8 | 2 | 5 | 24
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Prior Atorvastatin Use or Using Oral Atorvastatin [Count of Participants; unit: Participants]
  Prior Atorvastatin Use or Using Oral Atorvastatin | 6 | 4 | 1 | 5 | 16
  Prior Statin Other than Atorvastatin Use | 1 | 1 | 0 | 0 | 2
  No Prior Statin Use | 7 | 9 | 1 | 5 | 22

OUTCOME MEASURES:

1. Primary Outcome: Efficacy, Number of Participants With Day 15 LDL-C Less Than or Equal to 125% of Baseline LDL-C
Description: LDL-C levels were measured prior to and at the end of the 15 day treatment period to quantify the percent baseline LDL-C at 15 days. Efficacy is defined as eleven or more subjects in a dosing cohort with a Day 15 LDL-C not more than 125% of their baseline.
Time Frame: Baseline, 15 Days
Population: Efficacy Population: A completed group of subjects that 1) finished the two-week treatment period, 2) provided a Day 15 LDL-C level, and 3) took the final targeted dose for that cohort comprised the four efficacy populations.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 11 | 13 | 2 | 9
Participants | 9 | 9 | 1 | 7

2. Secondary Outcome: Efficacy, Number of Participants With Day 15 HDL-C More Than or Equal to 75% Baseline HDL-C
Description: HDL-C levels were measured prior to and at the end of the 15 day treatment period to quantify the percent baseline HDL-C at 15 days. Efficacy is defined as eleven or more subjects in a dosing cohort with a Day 15 HDL-C not less than 75% of their baseline.
Time Frame: Baseline, 15 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 11 | 13 | 2 | 9
Participants | 11 | 13 | 1 | 9

3. Secondary Outcome: Change in Baseline LDL-C Concentration
Description: Mean change in LDL-C (mg/dL) from baseline at Day 15
Time Frame: Baseline, 15 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 11 | 13 | 2 | 9
mg/dL | 12.36 (14.740) | 2.62 (34.844) | 27.50 (14.849) | 11.22 (13.283)

4. Secondary Outcome: Cmax IV
Description: The maximum serum concentration of atorvastatin and the 2- and 4-hydroxy active metabolites following an intravenous injection to a patient at steady-state.
Time Frame: 3 to 7 minutes, 0.5h, 1h 2h, 4h, 6h, 8h, 24h post-dose
Population: Pharmacokinetic Population: All subjects in the Efficacy Population who had no major protocol deviations and who had sufficient plasma atorvastatin concentration data for reliable estimates of the key PK variables for each of the four baseline cohorts.
Measure: Mean (Standard Deviation); unit: mg/mL
Groups:
- Cohort 1: Subjects taking 10 mg of oral atorvastatin daily at baseline will take targeted daily intravenous dose of 2 or 2.5 mg of atorvastatin injection for 15 days.
  Atorvastatin injection: statin (i.e., 3-hydroxy-3-methylglutaryl-coenzyme A (HMG-CoA) reductase inhibitor) for injection
- Cohort 2: Subjects taking 20 mg of oral atorvastatin daily at baseline will take targeted daily intravenous dose of 4 or 5 mg of atorvastatin injection for 15 days.
  Atorvastatin injection: statin (i.e., 3-hydroxy-3-methylglutaryl-coenzyme A (HMG-CoA) reductase inhibitor) for injection
- Cohort 3: Subjects taking 40 mg of oral atorvastatin daily at baseline will take targeted daily intravenous dose of 10 mg of atorvastatin injection for 15 days.
  Atorvastatin injection: statin (i.e., 3-hydroxy-3-methylglutaryl-coenzyme A (HMG-CoA) reductase inhibitor) for injection
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 11 | 13 | 2
mg/mL
  Atorvastatin | 284.33 (189.540) | 830.34 (1141.919) | 507.50 (443.456)
  2-Hydroxy Atorvastatin | 0.40 (0.87) | 1.23 (0.450) | 3.23 (1.987)
  4-Hydroxy Atorvastatin | 0.24 (0) | 0.30 (0.163) | 0.75 (0.370)

5. Secondary Outcome: Tmax IV
Description: The time to maximum concentration of atorvastatin and the 2- and 4-hydroxy active metabolites following an intravenous injection to a patient at steady-state.
Time Frame: 3 to 7 minutes, 0.5h, 1h 2h, 4h, 6h, 8h, 24h post-dose
Population: as for outcome 4
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 11 | 13 | 2
hours
  Atorvastatin | 0.08 [0.0 to 0.5] | 0.08 [0.0 to 0.5] | 0.15 [0.1 to 0.2]
  2-Hydroxy Atorvastatin | 6.00 [6.0 to 8.0] | 6.0 [2.0 to 8.0] | 5.00 [4.0 to 6.0]
  4-Hydroxy Atorvastatin | 0.08 [0.0 to 0.1] | 6.0 [0.0 to 8.0] | 8.0 [8.0 to 8.0]

6. Secondary Outcome: AUC 0-24
Description: The AUC 0-24 of atorvastatin and the 2- and 4-hydroxy active metabolites following an intravenous injection to a patient at steady-state.
Time Frame: 3 to 7 minutes, 0.5h, 1h 2h, 4h, 6h, 8h, 24h post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 11 | 13 | 2
ng*hr/mL
  Atorvastatin | 72.12 (31.216) | 137.04 (134.608) | 212.00 (89.095)
  2-Hydroxy Atorvastatin | 3.35 (2.603) | 16.76 (6.283) | 49.20 (26.698)
  4-Hydroxy Atorvastatin | NA (NA) — Values are below the level of detection | 5.45 (3.691) | 12.65 (5.303)

7. Secondary Outcome: AUC Inf
Description: The AUCinf of atorvastatin following an intravenous injection to a patient at steady-state.
Time Frame: 3 to 7 minutes, 0.5h, 1h 2h, 4h, 6h, 8h, 24h post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 11 | 13 | 2
ng*hr/mL | 72.19 (31.196) | 167.32 (138.099) | 217.00 (89.095)

8. Secondary Outcome: VDss
Description: The volume of distribution at steady state of atorvastatin following an intravenous injection to a patient.
Time Frame: 3 to 7 minutes, 0.5h, 1h 2h, 4h, 6h, 8h, 24h post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 11 | 13 | 2
liter | 71.86 (81.475) | 135.53 (145.579) | 182.85 (140.219)

9. Secondary Outcome: t 1/2
Description: The half-life of atorvastatin following an intravenous injection to a patient at a steady state.
Time Frame: 3 to 7 minutes, 0.5h, 1h 2h, 4h, 6h, 8h, 24h post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 11 | 13 | 2
hours | 4.79 (4.311) | 6.22 (1.884) | 6.38 (0.085)

ADVERSE EVENTS:
Time Frame: 15 days
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/2 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/2 | 0/10
Other Adverse Events (participants affected / at risk) | 4/14 | 1/14 | 1/2 | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=14) | Cohort 2 (N=14) | Cohort 3 (N=2) | Cohort 4 (N=10)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT03611010/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-10): https://cdn.clinicaltrials.gov/large-docs/10/NCT03611010/SAP_001.pdf